CLINICAL TRIAL: NCT05029258
Title: Biomarkers for Clinical Hypoxia Evaluation in Cervical Cancer
Acronym: Bio-CHECC
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ananya Choudhury, Professor in Clinical Oncology, Principal Investigator, University of Manchester
Other Study IDs: 20_DOG01_181
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer
Keywords: Hypoxia; Radiotherapy; Gene expression; Imaging
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hypoxia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy specimens retained
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Locally advanced cervical cancer patients treated with standard of care chemoradiation
  Interventions: Procedure: Biopsy of tumour; Diagnostic Test: MRI scans

INTERVENTIONS:
Procedure: Biopsy of tumour — Cervical tumour biopsy during treatment. This will be used for gene expression (RNA) analysis against a hypoxia associated gene signature.
Diagnostic Test: MRI scans — Multiple magnetic resonance imaging (MRI) scans before and during treatment using oxygen enhanced (OE) / tissues oxygen level dependent (TOLD) sequence

SUMMARY:
Patients with locally advanced cervical cancer (LACC) are primarily treated with radiotherapy +/- chemotherapy however 5-year survival rates are <60% with significant treatment toxicity. Hypoxia is a well-known radioresistant component of solid tumours such as cervical cancer and hypoxia modification therapies have demonstrated immense promise in treating such tumours. A major factor in determining a successful outcome with hypoxia modification is appropriate patient selection as it is hypoxic tumours that receive the most benefit from hypoxia modifying therapies. To date there is no validated hypoxia biomarker to stratify patients for therapy in cervical cancer in clinical use. This project offers a unique opportunity to examine both genetic and imaging biomarkers to optimise patient stratification when receiving curative radiotherapy for cervical cancer.

ELIGIBILITY:
Inclusion criteria:

* Patients must have a histologically confirmed diagnosis of cervical cancer
* Diagnostic/pre-treatment biopsy available
* Patients must be suitable for standard radiotherapy and brachytherapy
* Age greater than or equal to 18 years; no upper age limit
* Performance status - ECOG 0-2 (Refer to appendix 1)
* Women of childbearing age MUST have a negative pregnancy test prior to study entry and be using an adequate contraception method
* Before participant registration, written informed consent must be given according to GCP and national regulations.

Exclusion criteria:

* Participants deemed unsuitable for a biopsy (during or following radiotherapy) in the opinion of the treating oncologist.
* Patients with cardiac pacemakers, cochlear implants, intraocular foreign bodies or any other MR contraindication
* Patients with a hip replacement
* Patients with a known history of allergic reaction to gadolinium-based contrast agent
* Any contraindications to Hyoscine Butylbromide (Buscopan)
* Any patient taking ACE inhibitors. These should be stopped/substituted or they are a contraindication.
* Evidence of impaired renal function (eGFR <15 ml/min)
* Any evidence of severe or uncontrolled systemic diseases which, in the view of the investigator, makes it undesirable for the patient to participate in the study
* Evidence of significant clinical disorder or laboratory finding which, in the opinion of the investigator makes it undesirable for the patient to participate in the study
* Any other serious uncontrolled medical conditions
* Clinical evidence of metastatic disease
* Any pregnant or lactating woman
* Any patient with a medical or psychiatric condition that impairs their ability to give informed consent
* Any patient who is currently involved in, or who has recently been involved in other research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological sex based disease
Study Population: Locally advanced cervical cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
MRI derived hypoxia scores on 20 participants | 2 years
  20 patients will undergo functional imaging (hypoxia MRI) at baseline. Following this, serial measurements will be taken on a weekly basis during the first 5 weeks of chemoradiation. The imaging and biopsy cohorts are the same.
Gene signature derived hypoxia scores on the same 20 participants. | 2 years
  Investigators will collect paired biopsies at diagnosis and at brachytherapy in 20 locally advanced cervical cancer patients. The imaging and biopsy cohorts are the same.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No